CLINICAL TRIAL: NCT01434732
Title: A Randomized Controlled Trial of Umbilical Cord Milking Versus Immediate Cord Clamping on Systemic Blood Flow in Premature Infants
Brief Title: Effects of Milking the Umbilical Cord on Systemic Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Responsible Party: Principal Investigator, Anup Katheria, M.D., Director of Neonatal Research, Sharp HealthCare
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CORDMILK
Record Dates: First submitted 2011-06-03; First posted 2011-09-15 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Abnormal Vascular Flow
Keywords: Superior vena cava flow; umbilical cord milking; hemodynamics; systemic blood flow
MeSH Terms: interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Umbilical Cord Milking (Experimental): Umbilical Cord Milking involved milking the umbilical cord at birth.
  Interventions: Procedure: Umbilical Cord Milking
- Immediate Cord Clamping (Active Comparator): Umbilical cord is clamped soon after birth without any milking of the cord.
  Interventions: Procedure: Immediate Cord Clamping

INTERVENTIONS:
Procedure: Umbilical Cord Milking — UCM will be performed by the obstetric team by having the delivering obstetrician hold the infant below the mother's introitus at vaginal delivery or below the level of the incision at cesarean section and having the assistant (the second obstetrician) milk about 20 cm of umbilical cord over 2 seconds and repeating two additional times.
  Other Names: stripping the umbilical cord
  Arms: Umbilical Cord Milking
Procedure: Immediate Cord Clamping — The umbilical cord will be clamped soon after birth without any milking of the umbilical cord.
  Other Names: routine clamping of the umbilical cord
  Arms: Immediate Cord Clamping

SUMMARY:
Premature babies are at risk for bleeding in their brains, which can result in developmental delays or other neurological problems such as cerebral palsy. Clamping the baby's umbilical cord immediately after birth is standard, but delaying this procedure allows more of the baby's blood to move from the placenta into the baby and prevents head bleeds. However, a delay in clamping the umbilical cord is not usually done in very premature babies, because it would delay their treatment and they could get cold. Milking the umbilical cord is another way to give premature babies more of their own blood while avoiding a delay in treatment. Umbilical cord milking has been shown to improve blood pressure, decrease the need for blood transfusions, and increase the amount of urine made in the first few days of life.

DETAILED DESCRIPTION:
The aim of this study is to determine whether umbilical cord milking improves blood flow in premature babies, and thereby reduce the occurrence of neurological problems. The investigators predict that the blood flow measured by ultrasounds of the heart will be higher in babies who receive umbilical cord milking compared to those whose cords are clamped immediately. Secondly, the investigators predict that cord milking will improve blood volume, blood pressure, and urine output, and delay the need for blood transfusions.

This will be the first study to look at the effect that umbilical cord milking has on important measures of blood flow, which can predict bleeding in the head and subsequent developmental problems in very premature babies.

ELIGIBILITY:
Inclusion Criteria:

* infants < 32 weeks gestation

Exclusion Criteria:

* obstetrician's refusal to participate
* multiple gestations (if Di-Mo placentation) surrogate delivery
* parental desire for cord blood banking
* major congenital anomalies
* severe maternal illness
* placental abruption or previa
* ruptured uterus at delivery, or hemoperitoneum

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Superior Vena Cava Flow | 6 hours
  Researchers hypothesize that infants who receive umbilical cord milking (UCM) compared to infants who receive immediate cord clamping (ICC) will have higher SVC flow at 6 hours.

SECONDARY OUTCOMES:
Blood Pressure | 6 hours of life
  Researchers hypothesize that infants who receive umbilical cord milking (UCM) compared to infants who receive immediate cord clamping (ICC) will have higher blood pressures at 6 hours of life.
Neurodevelopmental Outcomes | between 18 and 36 months of life
  Researchers hypothesize that infants who receive umbilical cord milking (UCM) compared to infants who receive immediate cord clamping (ICC) will have improved neurodevelopmental outcomes. Neurodevelopmental follow-up data including cognitive, language, motor, social-emotional, and adaptive behavior composite scores from the Bayley Scales of Infant and Toddler Development (BSID-III) will be recorded when available. The presence of cerebral palsy, hearing and visual impairment will also be recorded when available.
number of blood transfusions | 36 weeks corrected gestational age
  Researchers hypothesize that infants who receive umbilical cord milking (UCM) compared to infants who receive immediate cord clamping (ICC) will have fewer blood transfusions at 36 weeks corrected gestational age.
Superior Vena Cava Flow | 18 hours of life
  Researchers hypothesize that infants who receive umbilical cord milking (UCM) compared to infants who receive immediate cord clamping (ICC) will have higher SVC flow at 18 hours.
Superior Vena Cava Flow | 30 hours of life
  Researchers hypothesize that infants who receive umbilical cord milking (UCM) compared to infants who receive immediate cord clamping (ICC) will have higher SVC flow at 30 hours.
Blood Pressure | at 18 hours of life
  Researchers hypothesize that infants who receive umbilical cord milking (UCM) compared to infants who receive immediate cord clamping (ICC) will have higher blood pressures at 18 hours of life.
Blood Pressure | 30 hours of life
  Researchers hypothesize that infants who receive umbilical cord milking (UCM) compared to infants who receive immediate cord clamping (ICC) will have higher blood pressures at 30 hours of life.

CONTACTS AND LOCATIONS:
Overall Officials: Anup C Katheria, M.D., Principal Investigator — UCSD
Locations (1):
- UCSD Medical Center, San Diego, California, United States

REFERENCES:
- [Derived] Katheria A, Garey D, Truong G, Akshoomoff N, Steen J, Maldonado M, Poeltler D, Harbert MJ, Vaucher YE, Finer N. A Randomized Clinical Trial of Umbilical Cord Milking vs Delayed Cord Clamping in Preterm Infants: Neurodevelopmental Outcomes at 22-26 Months of Corrected Age. J Pediatr. 2018 Mar;194:76-80. doi: 10.1016/j.jpeds.2017.10.037. Epub 2017 Dec 12. PMID 29246467
- [Derived] Katheria A, Blank D, Rich W, Finer N. Umbilical cord milking improves transition in premature infants at birth. PLoS One. 2014 Apr 7;9(4):e94085. doi: 10.1371/journal.pone.0094085. eCollection 2014. PMID 24709780
- [Derived] Katheria AC, Leone TA, Woelkers D, Garey DM, Rich W, Finer NN. The effects of umbilical cord milking on hemodynamics and neonatal outcomes in premature neonates. J Pediatr. 2014 May;164(5):1045-1050.e1. doi: 10.1016/j.jpeds.2014.01.024. Epub 2014 Feb 20. PMID 24560179